CLINICAL TRIAL: NCT02163837
Title: Effect of Rifaximine on Sleep Disorders in Patients Suffering From Hepatic Encephalopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Saint Pierre (Other)
Responsible Party: Principal Investigator, Marie Bruyneel, Chef de clinique, Centre Hospitalier Universitaire Saint Pierre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AK/14-02-14/4343
Record Dates: First submitted 2014-06-06; First posted 2014-06-16 (Estimated); Results first posted 2019-04-09 (Actual); Last update posted 2019-05-01 (Actual); Status verified 2019-04

CONDITIONS: Hepatic Encephalopathy
Keywords: sleep quality; physical activity; daytime sleepiness; actigraphy; quality of life
MeSH Terms: conditions — Hepatic Encephalopathy; Sleep Initiation and Maintenance Disorders; Motor Activity; Disorders of Excessive Somnolence | interventions — Rifaximin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- rifaximine (Experimental)
  Interventions: Drug: rifaximine

INTERVENTIONS:
Drug: rifaximine
  Other Names: Targaxan

SUMMARY:
Hepatic encephalopathy is responsible for sleep disturbances and daytime sleepiness. The purpose of our study is to assess sleep quality, quantity, sleep schemes and physical activity in patients suffering from HE, before and after a 2 weeks treatment with rifaximine, which is currently given to lower blood ammoniac levels.

DETAILED DESCRIPTION:
Hepatic encephalopathy (HE) is a complex neuropsychiatric syndrome related to chronic/acute hepatic failure. Sleep architecture is disturbed in this syndrome, and patients complain mainly of excessive daytime sleepiness and sleep disturbances. Hypothesis to explain these symptoms is, among others, disturbed melatonin metabolism. Few studies have been conducted in order to study sleep disorders during HE, and effect of treatment is unknown. Recently, rifaximine, an oral broad spectrum antibiotic, have been proved to decrease ammoniac production in patients with HE. The purpose of our study is to assess sleep quality, quantity, sleep schemes and physical activity in patients suffering from HE, before and after a 2 weeks treatment with rifaximine.

ELIGIBILITY:
Inclusion Criteria:

* >18y hepatic encephalopathy: positive Conn score

Exclusion Criteria:

* <18y pregnancy inability to fulfil questionnaires acute infection unstable clinical condition bone or articular disease resulting in significant disability

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2014-03; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marie Bruyneel, MD, Principal Investigator — CHU St Pierre
Locations (1):
- CHU St Pierre, Brussels, Belgium

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: all participants of this single arm study were actively enrolled
Groups:
- Rifaximine: rifaximine was given to all included patients after one week of assesment of sleep disturbances by polysomnography, actigraphy and questionnaires
Period: Before Rifaximin
Arm/Group | Rifaximine
Started | 15
Completed | 15
Not Completed | 0
Period: Day 28 of Rifaximin Treatment
Arm/Group | Rifaximine
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Rifaximine
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 57 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 9

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Slow Wave Sleep and REM Sleep
Description: sum of percentage of sleep spent in slow wave sleep and REM sleep during sleep per 24h ; assessed by 24-h polysomnography
Time Frame: 28 days
Measure: Mean (Standard Deviation); unit: percentage of total sleep time per 24h
Groups:
- Rifaximine: rifaximine
Arm/Group | Rifaximine
Number analyzed (Participants) | 15
percentage of total sleep time per 24h | 56 (16)

2. Secondary Outcome: Sleep Efficiency
Description: total sleep time/ time spent in bed per 24h, expressed in percentage of time spent in bed, assessed by actigraphy
Time Frame: 28 days
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Rifaximine
Number analyzed (Participants) | 15
percentage | 75 (7)

3. Other Pre Specified Outcome: Quality of Sleep
Description: assessed by Pittsburgh sleep quality index questionnaire (PSQI). Values: 0 to 21. 21= worse sleep quality
Time Frame: 28 days
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rifaximine
Number analyzed (Participants) | 15
units on a scale | 9 (5)

4. Other Pre Specified Outcome: Total Sleep Time
Description: total sleep time/ 24h, measured in minutes, by actigraphy
Time Frame: 28 days
Measure: Median (Full Range); unit: minutes
Arm/Group | Rifaximine
Number analyzed (Participants) | 15
minutes | 446 [53 to 701]

5. Other Pre Specified Outcome: Number of Steps Walked Daily
Description: number of steps walked daily assessed by actigraphy (measure of physical activity)
Time Frame: 28 days
Measure: Median (Full Range); unit: steps per day
Arm/Group | Rifaximine
Number analyzed (Participants) | 15
steps per day | 905 [56 to 5498]
Statistical Analysis 1: Comparison: Rifaximine; Mc Nemar symetry test for repeated measures and paired t-tests as appropriated; Test type: Superiority — the study was exploratory, the number of patients included was not calculated; p < 0.05, McNemar

ADVERSE EVENTS:
Time Frame: 28 days
Arm/Group | Rifaximine
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No